CLINICAL TRIAL: NCT04555616
Title: Environmental Design for Behavioral Regulation in People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth K Rhodus (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Elizabeth K Rhodus, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61291; T32AG057461 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease
Keywords: environment; Occupational therapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Placebo Comparator): Alzheimer's disease patients and caregivers.
  Interventions: Behavioral: Placebo
- Standard Environmental Design (Experimental): Alzheimer's disease patients and caregivers.
  Interventions: Behavioral: Standard Environmental Design
- Individualized Environmental Design Protocol (Experimental): Alzheimer's disease patients and caregivers.
  Interventions: Behavioral: Individual Environmental Design

INTERVENTIONS:
Behavioral: Standard Environmental Design — Participants' caregivers will receive set script of physical environmental modifications (i.e., declutter living space, reduce background noise, increase natural light), and social environment training script will include caregiving techniques: training for calming demeanor (emotional contagion), needs-driven care to decrease behavioral disruption, and accepting and accommodating approach to behavioral disruption. A pre-selected sensory stimulation kit will be provided to each participants' caregiver for administration throughout the day.
  Arms: Standard Environmental Design
Behavioral: Individual Environmental Design — Participants' caregivers will receive set script of physical environmental modifications and social environment training script in a standard protocol. Following initial assessments, individualized sensory stimulation kits will be developed using subjects' preferred sensory stimuli (as determined by the Adult Sensory Profile assessment and informant report) and will be provided via caregiver administration throughout the day to promote maintained behavioral regulation.
  Arms: Individualized Environmental Design Protocol
Behavioral: Placebo — Participants' caregivers will receive a set script of placebo modifications.
  Arms: Control Group

SUMMARY:
Individuals with dementia present with changes in behaviors throughout the continuum of cognitive decline. Environmental features may be influential in behavioral regulation. The purpose of this study is to assess the feasibility of environmental design protocols in older adults with dementia and their caregivers. Thirty subjects with moderate to severe Alzheimer's disease as primary dementia type, and their caregivers, will be randomly assigned to one of three arms: standard care; standard environmental design protocol; or personalized environmental design protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 21-90, inclusive.
* Living at home in the community with one primary caregiver.
* Diagnosis of Alzheimer's disease as primary dementia type of moderate to severe stages
* Stable medical condition for one month prior to screening visit
* Stable medications for 4 weeks prior to screening visit
* Caregiver report of challenges related to behaviors within 4 weeks of study enrollment
* Caregiver willing to participant throughout duration of study

Exclusion Criteria:

* Unstable medical conditions for 3 months prior to screening
* Wheelchair or bed bound.
* Residence in skilled nursing facility or facility-based care.
* Skin lesions or skin abnormalities throughout upper extremities.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Jicha, MD-PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentcuky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals diagnosed with Alzheimer's disease (Clinical Dementia Rating Scale [CDR] score of 1.0+) living in the community with caregiver-identified behavioral disturbance were recruited from the UK Alzheimer's Disease Research Center (UK ADRC)
Pre-assignment Details: Of 96 patient-caregiver dyads, 60 dyads were excluded (52 did not meet inclusion criteria; 4 declined to participate; 10 for other reasons.) Patients and their caregivers were enrolled as dyads. 30 dyads were randomized (10 to control, 10 to Standardized, 10 to Individualized) and 25 dyads completed the study.
Period: Overall Study
Arm/Group | Control Group | Standard Environmental Design | Individualized Environmental Design Protocol
Started (All numbers in this table represent dyads. One dyad is patient and their caregiver (total participants = 2 per dyad).) | 10 | 10 | 10
Completed (2 deaths report "patient" death.) | 7 | 9 | 9
Not Completed | 3 | 1 | 1
Not completed — Death | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Standard Environmental Design | Individualized Environmental Design Protocol | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Numbers of participants analyzed differ to drop of from study prior to study completion.
  years
    PLWD: number analyzed (Participants) | 6 | 7 | 9 | 22
    PLWD | 77.2 (7.4) | 84.3 (5.4) | 73.3 (7.1) | 77.9 (7.9)
    Caregiver: number analyzed (Participants) | 6 | 7 | 9 | 22
    Caregiver | 69.5 (14.0) | 67.7 (11.6) | 69.7 (11.7) | 69.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  PLWD: Female | 6 | 7 | 8 | 21
  PLWD: Male | 4 | 3 | 2 | 9
  Caregiver: Female | 9 | 8 | 2 | 19
  Caregiver: Male | 1 | 2 | 8 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  PLWD: American Indian or Alaska Native | 0 | 0 | 0 | 0
  PLWD: Asian | 0 | 0 | 0 | 0
  PLWD: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  PLWD: Black or African American | 1 | 0 | 0 | 1
  PLWD: White | 9 | 10 | 10 | 29
  PLWD: More than one race | 0 | 0 | 0 | 0
  PLWD: Unknown or Not Reported | 0 | 0 | 0 | 0
  Caregiver: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Caregiver: Asian | 0 | 0 | 0 | 0
  Caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Caregiver: Black or African American | 1 | 0 | 0 | 1
  Caregiver: White | 9 | 10 | 10 | 29
  Caregiver: More than one race | 0 | 0 | 0 | 0
  Caregiver: Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Education [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: Numbers of participants analyzed differ to drop of from study prior to study completion.
  years
    PLWD: number analyzed (Participants) | 7 | 7 | 9 | 23
    PLWD | 14.7 (3.2) | 14.6 (2.1) | 15.6 (2.0) | 15.0 (2.4)
    Caregiver: number analyzed (Participants) | 7 | 8 | 10 | 25
    Caregiver | 15.3 (2.5) | 16.3 (1.6) | 17.0 (2.4) | 16.3 (2.2)
Length of Caregiving Relationship [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: Numbers of participants analyzed differ to drop of from study prior to study completion.
  years
    number analyzed (Participants) | 7 | 5 | 8 | 20
    (all) | 3.7 (3.5) | 3.3 (2.9) | 5.6 (3.9) | 4.4 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Adherence
Description: Percentage of participants who had 75% adherence to the protocol based on visits and journals.
Time Frame: 6 weeks
Population: Difference of success rates among participants
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Standard Environmental Design | Individualized Environmental Design Protocol
Number analyzed (Participants) | 10 | 10 | 10
Participants | 2 | 6 | 7
Statistical Analysis 1: Comparison: Control Group vs Standard Environmental Design vs Individualized Environmental Design Protocol; Primary outcome analyzed via success rates among groups; Test type: Other; p = 0.12, Fisher Exact

2. Secondary Outcome: Change in Occupational Performance
Description: Occupational performance will be measured using the Canadian Occupational Performance Measure (COPM) at baseline, post-intervention and the 4-week follow up. Scores range from 0-10; higher scores indicate (increased) occupational performance.
Time Frame: 10 weeks (at baseline, 6 weeks and the 4 week follow up)
Population: Discontinued Intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Standard Environmental Design | Individualized Environmental Design Protocol
Number analyzed (Participants) | 7 | 7 | 8
score on a scale
  Baseline | 4.6 (0.4) | 3.6 (0.8) | 4.4 (0.8)
  Post Intervention: number analyzed (Participants) | 3 | 6 | 8
  Post Intervention | 4.6 (1.6) | 6.1 (1.1) | 6.6 (0.9)
  4-week follow up | 5 (1.4) | 5.2 (2.6) | 6.4 (2.6)

3. Secondary Outcome: Change in Behavior
Description: Behavior will be measured using the Neuropsychiatric Inventory (NPI-Q) at baseline, post-intervention and the 4-week follow up. Scores range from 1-36; higher scores indicate higher behavior severity.
Time Frame: 10 weeks (at baseline, 6 weeks and the 4 week follow up)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Standard Environmental Design | Individualized Environmental Design Protocol
Number analyzed (Participants) | 6 | 6 | 7
score on a scale
  Baseline | 13.3 (2.3) | 9.8 (2.8) | 10.3 (1.7)
  Post-Intervention | 8.9 (2.5) | 10.8 (1.9) | 8.4 (1.7)
  4-week follow up | 5.4 (2.7) | 5.5 (3.0) | 5.8 (3.7)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Mortality and Adverse Events were not monitored/collected for caregivers.
Arm/Group | Control Group | Standard Environmental Design | Individualized Environmental Design Protocol
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT04555616/Prot_SAP_ICF_001.pdf